CLINICAL TRIAL: NCT04889755
Title: SibACCESS: Developing a Telehealth Intervention to Address Unmet Psychosocial Needs of Siblings of Children With Cancer
Acronym: R03 CA259898
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Boston University Charles River Campus (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 5870E; R03CA259898 (NIH)
Record Dates: First submitted 2021-05-11; First posted 2021-05-17 (Actual); Results first posted 2025-02-17 (Actual); Last update posted 2025-02-17 (Actual); Status verified 2025-01

CONDITIONS: Siblings; Childhood Cancer; Pediatric Cancer; Posttraumatic Stress Disorder
MeSH Terms: conditions — Neoplasms; Stress Disorders, Post-Traumatic | interventions — Coping Skills

STUDY DESIGN:
Intervention Model Description: Parent Pre-session: Webinar on Supporting Siblings Session 1 (Sibling Group): Program Introduction Session 2 (Sibling Group): Understanding Emotions Session 3 (Sibling Group): Adaptive Thinking Session 4 (Sibling Group): Sitting with Emotions Session 5 (Sibling Group): Avoidance vs. Sitting with Emotions Sessions 6 (Sibling Individual): Telling Your Story Session 7 (Sibling Group): Keeping up with Skills Session 8 (Parent Individual): Parent/caregiver Check-In Session 9 (Sibling Group): Wrap-Up
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- SibACCESS (Other): This is a single-arm trial of a group-based, posttraumatic stress intervention for adolescent siblings of children with cancer. The intervention includes a parent educational webinar, seven group sibling sessions, one individual parent session, and one individual sibling session.
  Interventions: Behavioral: SibACCESS

INTERVENTIONS:
Behavioral: SibACCESS — The primary goal of the SibACCESS program is to increase siblings' exposure to and opportunity to process cancer-related cues to decrease onset or intensification of posttraumatic stress. The program is focused on siblings, with a brief parent education component. Parents will receive psychoeducation and brief skills training to support siblings enrolled in the program. Siblings will participate in 7 group sessions and one individual session in which they will learn skills and strategies to confront information about cancer and tolerate uncomfortable thoughts and feelings related to cancer, and thereby reduce avoidance of cancer-related emotions.
  Other Names: SibACCESS (Acceptance, Coping, Communication, Engagement, and Social Support)

SUMMARY:
This study aims to address barriers to psychosocial care for siblings of children with cancer by piloting a group-based telehealth program for adolescent siblings of youth with cancer. The pilot trial will be preceded by a treatment development stage during which study staff will interview English- and Spanish-speaking families and psychosocial providers to assess preferences for program content, format, timing, and cultural feasibility and acceptability, while considering ideas to minimize participation barriers. Information from interviews will inform any revisions to the proposed pilot program. Then, the new SibACCESS program will be tested with a small group of families located in Massachusetts, Delaware, or Rhode Island using video-teleconferencing technology. Families will complete exit interviews to assess program acceptability and perceived benefits.

DETAILED DESCRIPTION:
Background:

Prolonged, complicated, and intensive pediatric cancer treatment regimens challenge and disrupt the entire family. Siblings of youth with cancer are a psychosocially at-risk and underserved group. Siblings frequently report strong negative emotions, disruptions to family life, poorer academic functioning, more school absenteeism (school-aged siblings), and riskier health behaviors and poorer health outcomes than comparisons (adult siblings). Approximately one-quarter of siblings meet diagnostic criteria for cancer-related posttraumatic stress disorders. Outcomes are worse for siblings from under-represented minority groups and those with fewer socioeconomic resources. Additionally, siblings report low social support and indicate a strong desire to connect with other siblings. The need for sibling support is well established, as outlined in the recently developed evidence- and consensus-based Standards for Psychosocial Care for Children with Cancer and Their Families. Unfortunately, the Sibling Standard is among those least likely to be met within pediatric oncology programs nationwide.

SibACCESS Program Description:

SibACCESS (Acceptance, Coping, Communication, Engagement, and Social Support) targets the proposed mechanisms of sibling difficulties. The primary goal is to increase siblings' exposure and opportunities to process cancer-related cues to decrease the onset or intensification of posttraumatic stress (PTS). Treatment targets include emotional acceptance, treatment involvement, family communication (via between-session assignments), and social support (fostered by the group format).

SibACCESS is based on acceptance-based cognitive-behavioral frameworks, drawing primarily on trauma-focused CBT (TF-CBT). TF-CBT is a structured, short-term treatment that incorporates cognitive-behavioral approaches to promote recovery from trauma. It is a logical starting point for the present study for multiple reasons: (a) TF-CBT was developed specifically for children and adolescents; parent participation is recommended but not required; (b) it has been tested in a group format and using telehealth; (c) it has demonstrated effectiveness across cultural groups; and (d) it is appropriate for youth who meet diagnostic criteria for PTSD and those with sub-clinical PTS. TF-CBT has not yet been evaluated in the context of childhood cancer and may require some adaptations. Thus, SibACCESS also includes skills from Dialectical and Behavioral Therapy (i.e., self-validation of emotions, mindfulness, radical acceptance) to better address distress tolerance and acceptance of the aspects of cancer that are beyond siblings' control.

SibACCESS sessions will be facilitated remotely using Zoom. The intervention includes one pre-recorded parent webinar, one brief orientation meeting (sibling and parent), seven weekly sibling group sessions, one individual sibling session, and one individual parent session. The 30-minute parent webinar will provide a program overview, psychoeducation, and brief skills training. Parents will be given "discussion starter" questions to facilitate communication throughout the program. Sibling group sessions are 75 minutes and will include an ice breaker, review of last week's homework (except first session), introduction of new topics, interactive practice of new skills, and assignment of home practice (except final session). Exposure to cancer-related emotions and cues will be emphasized throughout the program, including talking about cancer, confronting cancer-related thoughts and emotions, selecting several individualized cancer-related exposures, and crafting a sibling narrative.

ELIGIBILITY:
Inclusion Criteria:

* 2 or more children in the family (i.e., child with cancer and >1 sibling)

  * Sibling(s) and child with cancer each under the age of 18 at the time of cancer diagnosis
  * Sibling(s) can be biologically-related, step-siblings, foster-siblings, or adopted-siblings
* Parent and sibling(s) fluent in English
* Sibling(s) 12-17 years of age
* Sibling report of at least mild posttraumatic stress (score >11 on the Child Posttraumatic Stress Scale for DSM-5)
* Child with cancer must have received cancer diagnosis at least 3 months prior to the family's enrollment in the study

Exclusion Criteria:

* A cognitive impairment that would interfere with pilot program and interview completion (as reported by parent)
* Bereavement
* Significant externalizing behaviors that would interfere with group participation (as reported by parent)

Min Age: 12 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Enrollment: 6 (Actual)
Dates: Start 2023-02-01 (Actual); Primary Completion 2023-06-10 (Actual); Study Completion 2023-06-10 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Kristin A. Long, PhD, Principal Investigator — Boston University
Locations (1):
- Boston University, Boston, Massachusetts, United States

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Groups:
- SibACCESS (Sibling Participants); SibACCESS (Parent Participants): This is a single-arm trial of a group-based, posttraumatic stress intervention for adolescent siblings of children with cancer. The intervention includes a parent educational webinar, seven group sibling sessions, one individual parent session, and one individual sibling session.
  SibACCESS: The primary goal of the SibACCESS program is to increase siblings' exposure to and opportunity to process cancer-related cues to decrease onset or intensification of posttraumatic stress. The program is focused on siblings, with a brief parent education component. Parents will receive psychoeducation and brief skills training to support siblings enrolled in the program. Siblings will participate in 7 group sessions and one individual session in which they will learn skills and strategies to confront information about cancer and tolerate uncomfortable thoughts and feelings related to cancer, and thereby reduce avoidance of cancer-related emotions.
Period: Overall Study
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants)
Started | 3 | 3
Completed (Participants reflect 3 sibling-parent family dyads (i.e. each enrolled sibling participated alongside an enrolled parent from their family)) | 3 | 3
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: This number represents 3 family dyads (including one sibling of a child with cancer and one parent participant from the same family per dyad) to complete the SibACCESS intervention
Groups:
- Total: Total of all reporting groups
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants) | Total
Number analyzed (Participants) | 3 | 3 | 6
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 3 | 0 | 3
  Between 18 and 65 years | 0 | 3 | 3
  >=65 years | 0 | 0 | 0
Age, Continuous [Mean (Standard Deviation); unit: Years] | 14.0 (1) | 41.3 (7.0) | 27.7 (15.6)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 2 | 2
  Male | 3 | 1 | 4
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 0 | 1
  Not Hispanic or Latino | 2 | 3 | 5
  Unknown or Not Reported | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0
  Asian | 0 | 0 | 0
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0
  Black or African American | 0 | 1 | 1
  White | 2 | 2 | 4
  More than one race | 1 | 0 | 1
  Unknown or Not Reported | 0 | 0 | 0
Region of Enrollment [Number; unit: participants]
  United States | 3 | 3 | 6
Sibling Perception Questionnaire (SPQ) [Mean (Standard Deviation); unit: units on a scale] — The Sibling Perception Questionnaire (SPQ) evaluates group interventions for siblings and parents designed to increase sibling understanding of and adjustment to chronic illness and developmental disability (CI/DD). Present measure was adapted from Sahler & Carpenter (1989) and Lobato & Kao (2002) versions to reflect cancer-related topics and create a parent-report version. Siblings and parents completed Sibling-report and Parent-report versions respectively. Measure was scored by a total summation, scores may range from 18 to 72.
  *Higher scores reflect more negative sibling adjustment
  units on a scale | 25 (11.3) | 35 (7.8) | 30 (10.3)
Strengths & Difficulties Questionnaire (SDQ) [Mean (Standard Deviation); unit: units on a scale] — The Strengths & Difficulties Questionnaire (Goodman, 1997) is a 25-item measure of children's psychosocial adjustment. It has five scales: Emotional Symptoms, Conduct Symptoms, Hyperactivity/ Inattention Symptoms, Peer Relationship Problems, and Prosocial Behavior. Adapted versions were given to sibling (self-report) and parent (parent-report) participants. Measure was scored by a total summation reflecting total child difficulties, scores may range from 0-40.
  *Higher scores reflect worse child difficulties
  units on a scale | 16.3 (5.9) | 19.3 (1.2) | 17.8 (4.1)
Child PTSD Symptom Scale for DSM-5 [Mean (Standard Deviation); unit: units on a scale] — The Child PTSD Symptom Scale for DSM-5 (CPSS-V) [citation] is a 27-item measure of posttraumatic stress. Strong test-retest reliability, internal consistency, and convergent validity with other child PTSD measures have been established. This survey was administered only to sibling participants. Measure was scored by a total summation, scores may range from 0 to 80.
  *Higher scores reflect higher levels of post-traumatic stress symptoms Population: Survey was administered only to sibling participants
  units on a scale
    number analyzed (Participants) | 3 | 0 | 3
    (all) | 12.7 (4.7) |  | 12.7 (4.7)
Coping self-efficacy scale [Mean (Standard Deviation); unit: units on a scale] — The Coping self-efficacy scale (Chesney et. al, 2006) was used to assess participants' confidence in performing coping behaviors when faced with life challenges. This measure was only used with sibling participants. Measure was scored by a total summation, scores may range from 0 to 260.
  *Higher scores reflect higher levels of coping self-efficacy Population: Survey was administered only to sibling participants
  units on a scale
    number analyzed (Participants) | 3 | 0 | 3
    (all) | 173 (49) |  | 173 (49)
Emotional Avoidance Strategy Inventory For Adolescents [Mean (Standard Deviation); unit: units on a scale] — The Emotional Avoidance Strategy Inventory for Adolescents (Kennedy & Ehrenreich-May, 2017) is a 17-item measure of emotional avoidance with acceptable psychometrics. Measure was scored by a total summation, scores may range from 0-68.
  *Higher scores reflect higher emotional avoidance Population: Survey was administered only to sibling participants
  units on a scale
    number analyzed (Participants) | 3 | 0 | 3
    (all) | 24 (16.8) |  | 24 (16.8)
Perceived Filial Self-Efficacy Scale [Mean (Standard Deviation); unit: units on a scale] — The Perceived Filial Self-Efficacy Scale (PFSES) (Caprara et. al, 2004) is a 16-item measure that assess efficacy beliefs that family members hold about their role as spouse, parent, and child, as well as about the functioning of family as a holistic system. This survey was administered only to sibling participants. Measure was scored by a total summation, scores may range from 16 to 112.
  *Higher scores reflect better efficacy beliefs Population: Survey was administered only to sibling participants
  units on a scale
    number analyzed (Participants) | 3 | 0 | 3
    (all) | 53.3 (19.0) |  | 53.3 (19.0)
Sibling Cancer Needs Inventory (SCNI) [Mean (Standard Deviation); unit: units on a scale] — The Sibling Cancer Needs Inventory (SCNI) (Patterson et. al, 2014) is a 45 item measure that assesses psychosocial needs of siblings are established to assist in the provision of appropriate support. This survey was administered only to sibling participants. The overall SCNI score are determined by summing the responses to all items, giving a possible range of SCNI scores from 45 to 180.
  *Higher scores reflect higher sibling psychosocial needs Population: Survey was administered only to sibling participants
  units on a scale
    number analyzed (Participants) | 3 | 0 | 3
    (all) | 67.3 (11.6) |  | 67.3 (11.6)

OUTCOME MEASURES:

1. Primary Outcome: Child Posttraumatic Stress Disorder Symptom Scale for DSM-5
Description: The Child PTSD Symptom Scale for DSM-5 (CPSS-V) [citation] is a 27-item measure of posttraumatic stress. Strong test-retest reliability, internal consistency, and convergent validity with other child PTSD measures have been established. This survey was administered only to sibling participants. Measure was scored by a total summation, scores may range from 0 to 80.
  *Higher scores reflect higher levels of post-traumatic stress symptoms
Time Frame: Within 2 weeks post-intervention, data were collected over a period of up to 4 weeks
Population: Survey was administered only to sibling participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants)
Number analyzed (Participants) | 3 | 0
units on a scale | 15.3 (3.5) |

2. Secondary Outcome: Strengths & Difficulties Questionnaire (SDQ)
Description: The Strengths & Difficulties Questionnaire (Goodman, 1997) is a 25-item measure of children's psychosocial adjustment. It has five scales: Emotional Symptoms, Conduct Symptoms, Hyperactivity/ Inattention Symptoms, Peer Relationship Problems, and Prosocial Behavior. Adapted versions were given to sibling (self-report) and parent (parent-report) participants. Measure was scored by a total summation reflecting total child difficulties, scores may range from 0-40.
  *Higher scores reflect worse child difficulties
Time Frame: Within 2 weeks post-intervention, data were collected over a period of up to 4 weeks
Population: Both sibling and parent participants completed this measure. One parent was unable to complete post-intervention measures.
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants)
Number analyzed (Participants) | 3 | 2.
units on a scale | 16.3 (5.5) | 13.0 (2.8)

3. Secondary Outcome: Sibling Perception Questionnaire (SPQ)
Description: The Sibling Perception Questionnaire (SPQ) evaluates group interventions for siblings and parents designed to increase sibling understanding of and adjustment to chronic illness and developmental disability (CI/DD). Present measure was adapted from Sahler & Carpenter (1989) and Lobato & Kao (2002) versions to reflect cancer-related topics and create a parent-report version. Siblings and parents completed Sibling-report and Parent-report versions respectively. Measure was scored by a total summation, scores may range from 18 to 72.
  *Higher scores reflect more negative sibling adjustment
Time Frame: Within 2 weeks post-intervention, data were collected over a period of up to 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants)
Number analyzed (Participants) | 3 | 2
units on a scale | 24.7 (13.9) | 36.5 (6.4)

4. Secondary Outcome: Coping Self-efficacy Scale
Description: The Coping self-efficacy scale (Chesney et. al, 2006) was used to assess participants' confidence in performing coping behaviors when faced with life challenges. This measure was only used with sibling participants. Measure was scored by a total summation, scores may range from 0 to 260.
  *Higher scores reflect higher levels of coping self-efficacy
Time Frame: Within 2 weeks post-intervention, data were collected over a period of up to 4 weeks
Population: Survey was administered only to sibling participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants)
Number analyzed (Participants) | 3 | 0
units on a scale | 188.0 (46.0) |

5. Secondary Outcome: Emotional Avoidance Strategy Inventory For Adolescents
Description: The Emotional Avoidance Strategy Inventory for Adolescents (Kennedy & Ehrenreich-May, 2017) is a 17-item measure of emotional avoidance with acceptable psychometrics. Measure was scored by a total summation, scores may range from 0-68.
Time Frame: Within 2 weeks post-intervention, data were collected over a period of up to 4 weeks
Population: Survey was administered only to sibling participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants)
Number analyzed (Participants) | 3 | 0
units on a scale | 11.7 (12.0) |

6. Secondary Outcome: Perceived Filial Self-Efficacy Scale
Description: The Perceived Filial Self-Efficacy Scale (PFSES) (Caprara et. al, 2004) is a 16-item measure that assess efficacy beliefs that family members hold about their role as spouse, parent, and child, as well as about the functioning of family as a holistic system. This survey was administered only to sibling participants. Measure was scored by a total summation, scores may range from 16 to 112.
  *Higher scores reflect better efficacy beliefs
Time Frame: Within 2 weeks post-intervention, data were collected over a period of up to 4 weeks
Population: Survey was administered only to sibling participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants)
Number analyzed (Participants) | 3 | 0
units on a scale | 89.7 (16.0) |

7. Secondary Outcome: Sibling Cancer Needs Inventory (SCNI)
Description: The Sibling Cancer Needs Inventory (SCNI) (Patterson et. al, 2014) is a 45 item measure that assesses psychosocial needs of siblings are established to assist in the provision of appropriate support. This survey was administered only to sibling participants. The overall SCNI score are determined by summing the responses to all items, giving a possible range of SCNI scores from 45 to 180.
  *Higher scores reflect higher sibling psychosocial needs
Time Frame: Within 2 weeks post-intervention, data were collected over a period of up to 4 weeks
Population: Survey was administered only to sibling participants
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants)
Number analyzed (Participants) | 3 | 0
units on a scale | 68.7 (15.5) |

8. Secondary Outcome: Acceptability of Program
Description: Based from the Client Satisfaction Questionnaire (Roberts et. el, 1984), this measure assesses participants general acceptability of the SibACCESS intervention. Measure was scored by a total summation, scores may range from 0 to 52.
  *Higher scores reflect higher levels of acceptability
Time Frame: Within 2 weeks post-intervention, data were collected over a period of up to 4 weeks
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants)
Number analyzed (Participants) | 3 | 2
units on a scale | 40.0 (7.0) | 40.0 (11.3)

ADVERSE EVENTS:
Time Frame: Through study completion, an average of 4 months
Arm/Group | SibACCESS (Sibling Participants) | SibACCESS (Parent Participants)
All-Cause Mortality (participants affected / at risk) | 0/3 | 0/3
Serious Adverse Events (participants affected / at risk) | 0/3 | 0/3
Other Adverse Events (participants affected / at risk) | 0/3 | 0/3

LIMITATIONS AND CAVEATS:
The present study explores the greater development of a psychosocial intervention program for siblings of children with cancer. Above outcomes reflect data from a proof of concept trial (Phase 2) regarding the SibACCESS program, which was not designed to measure statistically significant results.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol (2024-03-31): https://cdn.clinicaltrials.gov/large-docs/55/NCT04889755/Prot_000.pdf